CLINICAL TRIAL: NCT00935116
Title: Effect of the Administration of Etoricoxib on Postoperative Pain and Quality of Recovery in Patients Undergoing Thyroid Surgery
Brief Title: Etoricoxib for Postoperative Pain After Thyroid Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Padre Hurtado (Other)
Responsible Party: Alejandro Recart, MD, Padre Hurtado General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AR001cl
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- etoricoxib (Active Comparator): G1 (CONTROL): Oral NSAID (diclofenac, three times a day) administrated pre-operatively and for 3 days after surgery.
  G2: Etoricoxib 120 mg, pre and post-operatively for 3 days after surgery
  Interventions: Drug: etoricoxib

INTERVENTIONS:
Drug: etoricoxib — G1 (CONTROL): Oral NSAID (diclofenac, three times a day) administrated pre-operatively and for 3 days after surgery.
  G2: Etoricoxib 120 mg, pre and post-operatively for 3 days after surgery

SUMMARY:
The purpose of the study is evaluate the analgesic efficacy and safety profile of the Cox-2 specific analgesic Etoricoxib (arcoxia®) when administrated pre and postoperatively for controlling pain in adult patients undergoing thyroid surgery. Patients will be followed up in the immediate postoperative period, during the first postoperative (POD) day and in POD 2, 3 and 7. It is expected that with the addition of Etoricoxib, patients will experience less pain during the overall postoperative period and also a better quality of recovery when compared with the traditional analgesic regimen.

ELIGIBILITY:
Inclusion Criteria:

* age >18 and <70 years
* body weight within normal ranges
* ability to understand the use of pain assessment scales and the PCA device

Exclusion Criteria:

* known allergy to any of the drugs utilized
* contraindication to opioid and non-opioid analgesic drugs
* a history of bleeding disorders, peptic ulceration or anticoagulant use within the last month
* pregnant or breast-feeding patients
* history of known or suspected drug abuse or patients who had taken NSAIDs within 24 h prior to surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Maximum pain scores during postoperative period | every 6 hours, 24hours,48hours,72hours.

SECONDARY OUTCOMES:
Total amount of rescue analgesics | 24hours, 48hours, 72hours.